CLINICAL TRIAL: NCT01769053
Title: International Multicenter Randomized Controlled Open Trial on Variable vs. Non-Variable Pressure Support for Weaning From Mechanical Ventilation
Brief Title: Variable Pressure Support Trial
Acronym: ViPS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Rate of recruitment
Sponsor: Technische Universität Dresden (Other)
Collaborators: Medical University of Vienna (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); University Hospital, Montpellier (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other); St Thomas' Hospital, London (Other); Hospital Sírio-Libânes, São Paulo, Brazil (Unknown); Hospital Copa D'Or, Rio de Janeiro, Brazil (Unknown); Hospital Universitari Sant Joan de Reus (Other); University of Kiel (Other); Fachkrankenhaus Coswig GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK235082012
Record Dates: First submitted 2012-12-18; First posted 2013-01-16 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Acute Lung Injury; Adult Respiratory Distress Syndrome; at Least 24 h of Controlled Mechanical Ventilation
Keywords: Acute Lung Injury; Adult Respiratory Distress Syndrome; Interactive Ventilatory Support; Positive-Pressure Respiration; Ventilator-Induced Lung Injury
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome; Ventilator-Induced Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Variable Ventilation (Active Comparator): Patients are ventilated with variable pressure support mode.
  Interventions: Other: Variable Ventilation
- Conventional (non-variable) Ventilation (No Intervention): Patients are ventilated with non-variable(conventional) pressure support ventilation mode.

INTERVENTIONS:
Other: Variable Ventilation
  Arms: Variable Ventilation

SUMMARY:
In 2008 a new ventilation strategy termed variable Pressure Support ventilation (PSV) was introduced, which is able to increase the variability of the respiratory pattern independent from the inspiratory effort. In experimental lung injury, variable PSV was found to improve gas exchange and decrease the inspiratory effort, while reducing alveolar edema and inflammatory infiltration compared to conventional(non-variable) PSV. Importantly, variable PSV reduced peak airway pressure and respiratory system elastance in a variability dependent manner.In addition, preliminary observations suggest that variable PSV can reduce the work of breathing and improve patient comfort, but it is not known whether this new ventilatory strategy is able to speed the weaning from mechanical ventilation.

Since variable PSV can reduce the mean pressure support, it may lead to a faster reduction of pressure support and, therefore, a shorter weaning period than conventional PSV.

The hypothesis of this study is that variable pressure support ventilation reduces the duration of mechanical ventilation to non-variable (conventional) pressure support ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Duration of controlled mechanical ventilation ≥ 24h
* Availability of a Infinity V500 ventilator (ready to use)
* Informed consent according to local regulations
* Temperature ≤ 39 °C
* Hemoglobin ≥ 6 g/dl
* PaO2/FIO2 ≥ 150 mmHg with positive end-expiratory pressure (PEEP) ≤16 cmH2O
* Ability to breath spontaneously

Exclusion Criteria:

* Participation in another interventional trial within the last four weeks before enrollment in this trial
* Peripheral neurological disease associated with impairment of the respiratory pump
* Muscular disease associated with impairment of the respiratory pump
* Instable thorax with paradoxical chest wall movement
* Planned surgery under general anesthesia within 72 hours
* Difficult airway/intubation
* Existing tracheotomy at ICU admission
* Expected survival < 72 hours
* Home mechanical ventilation or on chronic oxygen therapy
* Suspected pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2013-01; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Weaning time | From time of randomization until the time of successful extubation, estimated to be up to 30 days
  Weaning time defined as time from randomization to successful extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Gama de Abreu, Principal Investigator — Dresden University
Locations (1):
- Department of Anesthesiology and Intensive Care, Dresden University of Technology, Dresden, Germany

REFERENCES:
- [Derived] Kiss T, Guldner A, Bluth T, Uhlig C, Spieth PM, Markstaller K, Ullrich R, Jaber S, Santos JA, Mancebo J, Camporota L, Beale R, Schettino G, Saddy F, Vallverdu I, Wiedemann B, Koch T, Schultz MJ, Pelosi P, de Abreu MG. Rationale and study design of ViPS - variable pressure support for weaning from mechanical ventilation: study protocol for an international multicenter randomized controlled open trial. Trials. 2013 Oct 31;14:363. doi: 10.1186/1745-6215-14-363. PMID 24176188
- See also: Institution's and project's website — http://www.peg-dresden.de